CLINICAL TRIAL: NCT07336940
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Single and Multiple-Dose Escalation, and Food Effect Study of ENV-294 in Healthy Adult Participants With a Phase 1b Extension in Adults With Moderate-To-Severe Atopic Dermatitis
Brief Title: Study of ENV-294 in Healthy Adults and in Adults With Moderate-to-Severe Atopic Dermatitis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Enveda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENV-294-101
Record Dates: First submitted 2025-09-20; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label with once per day dosing (Experimental)
  Interventions: Drug: ENV-294 Capsule

INTERVENTIONS:
Drug: ENV-294 Capsule — ENV-294 formulated as 200mg capsules for oral administration will be used for this study.

SUMMARY:
The goal of this clinical trial is to learn about the safety and tolerability of ENV-294 in adults with moderate to severe atopic dermatitis. It may also learn about the changes ENV-294 may have on the severity of atopic dermatitis symptoms.

The main questions it will answer are:

* Is ENV-294 safe and well tolerated in adults with moderate to severe atopic dermatitis?
* Is there an impact on the severity of atopic dermatitis symptoms when participants take ENV-294? Researchers will review the atopic dermatitis present at the beginning of the study against the atopic dermatitis present at the end of the study.

Participants will:

* Take drug ENV-294 once every day for 28 days
* Visit the clinic weekly for 4 weeks for checkups and tests
* Keep a diary of their symptoms and when they took their study drug ENV-294

ELIGIBILITY:
Inclusion Criteria:

* Be male or female participants who are 18 to 75 years of age
* Have chronic AD (also known as atopic eczema) that was diagnosed at least 12 months prior to the first study visit
* Have a history of inadequate response or intolerance to topical corticosteroids or other topical treatments for used atopic dermatitis
* Have moderate-to-severe atopic dermatitis, at the first two study visits
* Use an emollient (except those containing urea) daily for at least 1 week prior to the first study visit and throughout the study

Exclusion Criteria:

* Have any uncontrolled current or recurrent concomitant illness (eg, hepatitis B surface antigen, hepatitis C virus, or other condition) that could affect the study drug, clinical or laboratory assessments, or could impact participant safety.
* Are using any medication (prescription or over-the-counter) that may interfere with the study product safety evaluations within 14-days prior to the second study visit.
* Have the presence of any concomitant skin conditions (eg, psoriasis, seborrheic dermatitis) or have large tattoos that would interfere with clinical assessment, evaluation of AD, or treatment response.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of ENV-294 when administered to adult participants with moderate-to-severe atopic dermatitis. | From enrollment through treatment and the final study visit at approximately day 42.
  Incidence and severity of adverse events, serious adverse events and adverse events leading to the discontinuation of treatment.
Incidence of abnormalities in clinical chemistry parameters as a measure of safety and tolerability of ENV-294. | Baseline through end of study at approximately Day 42.
  The number of participants with clinically significant abnormalities in clinical chemistry parameters will be assessed to evaluate safety and tolerability of multiple escalating doses of ENV-294.
To assess the safety and tolerability of ENV-294 when administered to adult participants with moderate-to-severe atopic dermatitis | From first dose through treatment and the final study visit at approximately day 42.
  Incidence of clinically significant changes in physical exam findings after ENV-294 administration.
Incidence of clinically significant changes in systolic blood pressure (mmHg) as a measure of safety and tolerability of ENV-294. | From first dose through treatment and the final study visit at approximately day 42.
  The number of participants with clinically significant increases or decreases in systolic blood pressure, measured in millimeters of mercury (mmHg), will be assessed to evaluate the safety and tolerability of ENV-294 in adults with moderate-to-severe atopic dermatitis.
Incidence of clinically significant changes in heart rate (beats per minute) measured by 12-lead ECG as a measure of safety and tolerability of ENV-294. | Baseline through treatment and the final study visit at approximately day 42.
  The number of participants with clinically significant changes in heart rate, measured in beats per minute from 12-lead ECG recordings, will be assessed to evaluate the cardiac safety and tolerability of ENV-294 in adults with moderate-to-severe atopic dermatitis.
Incidence of abnormalities in hematology parameters as a measure of safety and tolerability of ENV-294. | Baseline through the end of the study at approximately Day 42.
  The number of participants with clinically significant abnormalities in hematology parameters (e.g., hemoglobin, hematocrit, red blood cell count, white blood cell count, platelet count) will be assessed to evaluate safety and tolerability of multiple escalating doses of ENV-294.
Incidence of abnormalities in coagulation parameters as a measure of safety and tolerability of ENV-294. | Baseline through the end of the study at approximately Day 42.
  The number of participants with clinically significant abnormalities in coagulation parameters (e.g., PT, aPTT, INR) will be assessed to evaluate safety and tolerability of multiple escalating doses of ENV-294.
Incidence of abnormalities in urinalysis parameters as a measure of safety and tolerability of ENV-294. | Baseline through the end of the study at approximately Day 42.
  The number of participants with clinically significant abnormalities in urinalysis parameters (e.g., specific gravity, protein, glucose, blood, leukocytes) will be assessed to evaluate safety and tolerability of multiple escalating doses of ENV-294.
Incidence of clinically significant changes in diastolic blood pressure (mmHg) as a measure of safety and tolerability of ENV-294. | Baseline through treatment and the final study visit (approximately Day 42).
  The number of participants with clinically significant increases or decreases in diastolic blood pressure, measured in millimeters of mercury (mmHg), will be assessed to evaluate the safety and tolerability of ENV-294 in adults with moderate-to-severe atopic dermatitis.
Incidence of clinically significant changes in heart rate as a measure of safety and tolerability of ENV-294. | Baseline through treatment and the final study visit (approximately Day 42).
  The number of participants with clinically significant changes in heart rate (beats per minute) will be assessed to evaluate the safety and tolerability of ENV-294 in adults with moderate-to-severe atopic dermatitis.
Incidence of clinically significant changes in respiratory rate as a measure of safety and tolerability of ENV-294. | Baseline through treatment and the final study visit (approximately Day 42).
  The number of participants with clinically significant changes in respiratory rate (breaths per minute) will be assessed to evaluate the safety and tolerability of ENV-294 in adults with moderate-to-severe atopic dermatitis
Incidence of clinically significant changes in body temperature as a measure of safety and tolerability of ENV-294. | Baseline through treatment and the final study visit (approximately Day 42).
  The number of participants with clinically significant changes in body temperature (°C) will be assessed to evaluate the safety and tolerability of ENV-294 in adults with moderate-to-severe atopic dermatitis.
Incidence of clinically significant changes in RR interval (milliseconds) measured by 12-lead ECG as a measure of safety and tolerability of ENV-294. | Baseline through treatment and the final study visit (approximately Day 42).
  The number of participants with clinically significant changes in RR interval, measured in milliseconds (ms) from 12-lead ECG recordings, will be assessed to evaluate the cardiac safety and tolerability of ENV-294.
Incidence of clinically significant changes in PR interval (milliseconds) measured by 12-lead ECG as a measure of safety and tolerability of ENV-294. | Baseline through the end of the study at approximately Day 42.
  The number of participants with clinically significant changes in PR interval, measured in milliseconds (ms) from 12-lead ECG recordings, will be assessed to evaluate cardiac conduction safety of ENV-294.
Incidence of clinically significant changes in QRS duration (milliseconds) measured by 12-lead ECG as a measure of safety and tolerability of ENV-294. | Baseline through treatment and the final study visit (approximately Day 42).
  The number of participants with clinically significant changes in QRS duration, measured in milliseconds (ms) from 12-lead ECG recordings, will be assessed to evaluate cardiac conduction safety of ENV-294.
Incidence of clinically significant changes in QT interval (milliseconds) measured by 12-lead ECG as a measure of safety and tolerability of ENV-294. | Baseline through treatment and the final study visit (approximately Day 42).
  The number of participants with clinically significant changes in QT interval, measured in milliseconds (ms) from 12-lead ECG recordings, will be assessed to evaluate cardiac repolarization safety of ENV-294.
Incidence of clinically significant changes in QTc Bazett (milliseconds) measured by 12-lead ECG as a measure of safety and tolerability of ENV-294. | Baseline through treatment and the final study visit (approximately Day 42)
  The number of participants with clinically significant changes in QTc Bazett (QT corrected for heart rate using Bazett's formula), measured in milliseconds (ms), will be assessed to evaluate cardiac safety of ENV-294.
Incidence of clinically significant changes in QTc Fridericia (milliseconds) measured by 12-lead ECG as a measure of safety and tolerability of ENV-294. | From enrollment through treatment and the final study visit (approximately Day 42)
  The number of participants with clinically significant changes in QTc Fridericia (QT corrected for heart rate using Fridericia's formula), measured in milliseconds (ms), will be assessed to evaluate cardiac safety of ENV-294.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of ENV-294 | Pre and/or post-dose on days 1, 8, 15 and 28, and on day 42.
  Maximum observed plasma concentration (Cmax) of ENV-294 will be determined from plasma samples collected at scheduled time points following oral administration to evaluate pharmacokinetic properties.
Time to reach maximum plasma concentration (Tmax) of ENV-294 | Pre and/or post-dose on days 1, 8, 15 and 28, and on day 42.
  Time to reach maximum observed plasma concentration (Tmax) of ENV-294 will be determined from plasma concentrations measured at scheduled post-dose time points.
Area under the plasma concentration-time curve from time zero to 24 hours (AUC₀-₂₄h) of ENV-294 | Pre and/or post-dose on days 1, 8, 15 and 28, and on day 42.
  Area under the plasma concentration-time curve from time zero to 24 hours (AUC₀-₂₄h) will be calculated from measured plasma concentrations of ENV-294 to assess systemic drug exposure after multiple oral doses.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Skin Sciences, PLLC, Louisville, Kentucky
  - J & S Studies, College Station, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Virginia Dermatology & Skin Cancer Center, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Undecided